CLINICAL TRIAL: NCT01825941
Title: Diphenhydramine as Adjuvant Therapy for Acute Migraine. A Randomized Trial.
Brief Title: Diphenhydramine for Acute Migraine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Benjamin W. Friedman, MD, Associate professor of Emergency Medicine, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-02-071
Record Dates: First submitted 2013-04-02; First posted 2013-04-08 (Estimated); Results first posted 2018-06-08 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Migraine
Keywords: migraine; headache; metoclopramide; diphenhydramine
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Metoclopramide; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metoclopramide + Diphenhydramine (Active Comparator): Metoclopramide 10 milligrams + Diphenhydramine 50 milligrams, administered as an intravenous drip over 15 minutes
  Interventions: Drug: metoclopramide; Drug: diphenhydramine
- Metoclopramide + placebo (Placebo Comparator): Metoclopramide 10mg + placebo, administered intravenously over 15 minutes
  Interventions: Drug: metoclopramide; Drug: placebo

INTERVENTIONS:
Drug: metoclopramide — 10 milligrams, administered intravenously over 15 minutes
  Other Names: Reglan
Drug: diphenhydramine — 50 milligrams, administered intravenously over 15 minutes
  Other Names: Benadryl
  Arms: Metoclopramide + Diphenhydramine
Drug: placebo
  Arms: Metoclopramide + placebo

SUMMARY:
Parenteral diphenhydramine is commonly used as adjuvant therapy for acute migraine despite the fact that data supporting this practice do not exist. The investigators propose a randomized double blind study to test the hypothesis that 50mg of intravenous diphenhydramine, when added to standard migraine therapy, will result in a greater rate of sustained headache relief than standard migraine therapy alone. For this study, standard migraine therapy will be 10mg of intravenous metoclopramide. Sustained headache relief is defined as achieving a headache level of "mild" or "none" within two hours and maintaining a level of "mild" or "none" for 48 hours. Patients who present to the Montefiore emergency room (Bronx, NY) with an acute migraine will be approached for participation. They will be screened for medication contra-indications and non-migraine etiologies of headache. The study will be randomized. Assignment will be concealed. Participants and researchers will be blinded. Efficacy outcomes and adverse events will be assessed every half hour for two hours in the Emergency Department and by telephone 48 hours after medication administration. A sample size calculation, based on pilot data, revealed the need for 374 participants. An interim analysis will be performed after 200 participants have been enrolled with the goal of assessing for lack of conditional power.

ELIGIBILITY:
Inclusion Criteria:

* Acute migraine headache
* Present to our emergency room in the Bronx, NY for treatment of migraine headache

Exclusion Criteria:

* Temperature > 100.3 F
* Pheochromocytoma
* Seizure disorder
* Parkinson's disease
* Use of monoamine oxidase (MAO) inhibitors
* Use of anti-rejection transplant medications
* Use of potassium supplements
* Use of pramlintide

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 208 (Actual)
Dates: Start 2013-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin W Friedman, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Derived] Friedman BW, Cabral L, Adewunmi V, Solorzano C, Esses D, Bijur PE, Gallagher EJ. Diphenhydramine as Adjuvant Therapy for Acute Migraine: An Emergency Department-Based Randomized Clinical Trial. Ann Emerg Med. 2016 Jan;67(1):32-39.e3. doi: 10.1016/j.annemergmed.2015.07.495. Epub 2015 Aug 29. PMID 26320523

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol anticipated enrollment of around 400 participants, however Data Safety Monitoring Board recommended enrollment cut to approximately half
Groups:
- Metoclopramide + Placebo: Metoclopramide 10mg + placebo, administered intravenously over 15 minutes
  metoclopramide: 10 milligrams, administered intravenously over 15 minutes
  placebo
Period: Overall Study
Arm/Group | Metoclopramide + Diphenhydramine | Metoclopramide + Placebo
Started | 104 | 104
Completed | 100 | 103
Not Completed | 4 | 1
Not completed — Lost to Follow-up | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metoclopramide + Diphenhydramine | Metoclopramide + Placebo | Total
Number analyzed (Participants) | 104 | 104 | 208
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (11) | 36 (10) | 35 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 92 | 180
  Male | 16 | 12 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 104 | 104 | 208
Duration of headache Prior to Study [Median (Inter-Quartile Range); unit: Hours] | 72 [24 to 96] | 48 [16 to 72] | 48 [24 to 96]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sustained Headache Relief Assessed by Self-evaluation
Description: Sustained headache relief is defined as achieving a headache level of "mild" or "none" within two hours and maintaining a level of "mild" or "none" for 48 hours. Patient self-evaluated pain level is solicited every half hour for two hours in the Emergency Department and then by telephone 48 hours after discharge from emergency department
Time Frame: up to 2 hours in Emergency Department, 48 hours after discharge from Emergency Department
Measure: Count of Participants; unit: Participants
Arm/Group | Metoclopramide + Diphenhydramine | Metoclopramide + Placebo
Number analyzed (Participants) | 100 | 103
Participants | 40 | 38

ADVERSE EVENTS:
Arm/Group | Metoclopramide + Diphenhydramine | Metoclopramide + Placebo
All-Cause Mortality (participants affected / at risk) | 0/104 | 0/104
Serious Adverse Events (participants affected / at risk) | 0/104 | 0/103
Other Adverse Events (participants affected / at risk) | 25/104 | 21/104
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metoclopramide + Diphenhydramine (N=104) | Metoclopramide + Placebo (N=104)
Restlessness (Nervous system disorders) | 8 (8) | 7 (7)
Drowsy (Nervous system disorders) | 17 (17) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes